CLINICAL TRIAL: NCT02642081
Title: Non-steroidal Anti-inflammatory Drugs (NSAIDs) and Risk of Acute Kidney Injury in Patients With Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201511075RIND
Record Dates: First submitted 2015-12-17; First posted 2015-12-30 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure
Keywords: NSAIDs; Heart failure; Acute kidney injury
MeSH Terms: conditions — Heart Failure; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate whether non-steroidal anti-inflammatory drugs (NSAIDs) were associated with acute kidney injury (AKI) in patients with heart failure. In addition, the investigators would like to assess the risk of admission for acute decompensated heart failure following exposure to NSAIDs within 30 days.

ELIGIBILITY:
Inclusion criteria

1. Patient's age was more than 20 years old
2. Diagnosis of heart failure
3. With prescription of NSAIDs (only oral and intravenous form are included)

Exclusion criteria

1. With prescription of NSAIDs administered by topical use
2. Patient was pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with prescription of NSAIDs
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in serum creatinine at 1 month | Baseline and 1 month
  We collect not only patient's baseline serum creatinine level (defined as the median value of the previous-six-months serum creatinine), but also serum creatinine level on the detecting day (defined as the most recent day from index date we detecting the serum creatinine). Acute kidney injury is defined as the absolute increase in the serum creatinine concentration of ≥0.3 mg/dL from baseline; or a percentage increase in the serum creatinine concentration of ≥50 percent.

SECONDARY OUTCOMES:
Admission for acute decompensated heart failure | 1 month after exposure to NSAIDs

CONTACTS AND LOCATIONS:
Overall Officials: Chii-Ming Lee, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan